CLINICAL TRIAL: NCT07216222
Title: Intracranial Recording and Stimulation of the Human Hippocampal-Amygdala Circuit During Virtual Reality Fear Conditioning
Brief Title: K08 VR Fear Conditioning
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Duke University (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony Jang, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-24-6010; 1K08MH138741-01 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Anxiety and Fear; PTSD; Veteran
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All RNS Participants (Experimental): In this single-arm study, all participants will complete identical experimental conditions with simultaneous iEEG recordings (Recording Study) or iEEG stimulation (Stimulation Study).
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep brain stimulation via the Responsive Neurostimulator (RNS) device.

SUMMARY:
The goal of this clinical trial is to learn how people respond to fear-related experiences in a virtual reality (VR) environment. The study will also look at how brain activity and body responses are connected to learning and memory of fear. To do so, we recruit individuals who are already implanted with a Responsive Neurostimulator (RNS) device for the treatment of epilepsy. This research may help improve our understanding of anxiety disorders and how to better treat them in the future.

The main questions it aims to answer are: 1) How do people learn to associate certain cues in VR with feelings of fear or safety? 2) What brain and body responses happen during fear learning?

Participants will: 1) Wear a virtual reality headset and experience different environments and sounds, 2) Have their brain activity, heart rate, and sweating measured, and 3) Receive safe, mild electrical pulses through the RNS device during the study to help study fear learning. Participants will attend one or more study sessions, each lasting about 3-4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Female
* Between 18 and 70 years of age
* Adequate visual and auditory acuity to allow neuropsychological testing
* Have undergone surgical placement of NeuroPace RNS System for the treatment of epilepsy or post-traumatic stress disorder

Exclusion Criteria:

- History of traumatic brain injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Intracranial EEG activity | Baseline
  Power in the theta band (~3-12 Hz).
Skin conductance activity | Baseline
  Electrodermal response during the fear conditioning experiment, as quantified by changes in electrical conductance between electrodes placed on the palm.
Heart rate | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT07216222/Prot_SAP_000.pdf